CLINICAL TRIAL: NCT04220216
Title: A Pilot Study to Assess the Haymakers for Hope Fitness Program in Cancer Survivors
Brief Title: Pilot Study of the Haymakers for Hope Fitness Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID pandemic
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Haymakers for Hope (Unknown)
Responsible Party: Principal Investigator, Elizabeth O'Donnell, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-426
Record Dates: First submitted 2019-12-19; First posted 2020-01-07 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Cancer; Exercise Test; Fatigue; Mood; Quality of Life; Biomarkers
Keywords: Cancer; Exercise Test; Cardiopulmonary Exercise Test; Fatigue; Mood; Quality of Life; Biomarkers; Analysis, Survival
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- H4H fitness program (Experimental): The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.
  * Patients will attend the 16-week program of boxing conditioning.
  * This 16-week program will include supervised exercises designed to improve strength, flexibility, balance,and cardiopulmonary fitness.
  * There will be 4, 1-hour sessions each week per participant
  Interventions: Other: H4H fitness program

INTERVENTIONS:
Other: H4H fitness program — 4 weekly, 1 hour exercise sessions

SUMMARY:
This research study is assessing the effect of an exercise program on cancer survivors.

The exercise program is Haymakers for Hope 16-week exercise program

DETAILED DESCRIPTION:
This is a pilot study, it is the first time investigators are examining the effect of this exercise program on cancer survivors physical and emotional functioning. The exercise programs is based on the conditioning program used by boxers.- Haymakers for Hope 16-week exercise program

* The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.
* Participants will attend the 16-week program of boxing conditioning. It is expected that about 10 people will take part in this research study.

  * This 16 week will include supervised exercises designed to improve strength, flexibility, balance and cardiopulmonary fitness.
  * There will be 4 sessions of 1 hour each week for each of the 10 participants.
  * The program will be conducted at gymnasiums contracted with the H4H program and outcomes assessments at Massachusetts General Hospital and the gymnasiums..

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis excluding non-melanoma skin cancer
* Age ≥ 18 years
* ECOG performance status ≤1
* Medical clearance by treating clinician
* No known contraindications to moderate intensity exercise such as (but not limited to) brain metastases, serious or non-healing wound, peripheral neuropathy greater than or equal to Grade 3, or myocardial infarction within 1- year.
* Able to complete forms and understand instruction in English
* Willing and able to attend the H4H program for 16 weeks
* Willing and able to complete the baseline and follow-up visits at MGH
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Participants who have had surgery within 4 weeks prior to entering the study or those who have not recovered from adverse events due to surgery more than 4 weeks earlier.
* Blastic or lytic bone lesions
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Chest pain brought on by physical activity
* Pregnant women or women intending to become pregnant during the study period
* Presence of dementia or major psychiatric illness that would preclude participation in a group program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Rate of Attendance | 16 weeks
  Participants will be considered to have completed the fitness program if they attend at least 70% of the sessions
Rate of Completion | 16 weeks
  Feasibility will be demonstrated if ≥60% of participants complete the fitness program

SECONDARY OUTCOMES:
Change in cardiopulmonary fitness as assessed by the 6-minute walk test | 16 weeks
  summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences
Change in strength | 16 weeks
  summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences
Change in QOL as assessed by the Functional Assessment of Cancer Therapy - General | 16 weeks
  summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences
Change in psychological well-bring as assessed by the Ryff Psychological Well-Being Scale (Min score: 42, Max score: 252. A higher score indicating higher psychological well-being) | 16 weeks
  summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences
Change in fatigue as assessed by Functional Assessment of Chronic Illness Therapy - Fatigue | 16 weeks
  summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences
Change in sleep quality as assessed by the Rand Medical Outcome Survey (MOS) Sleep Scale (min score: 0; max score: 100. A higher core indicates more sleep problems) | 16 weeks
  summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences
Change in anxiety as assessed by Hospital Anxiety and Depression Scale (HADS) (min score: 0; max score: 21. A higher score indicates more anxiety) | 16 weeks
  summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences
Change in depression as assessed by Hospital Anxiety and Depression Scale (HADS) (min score: 0; max score: 21. A higher score indicates more depression) | 16 weeks
  summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences
Change in body composition as assessed by change in total lean mass, extremity lean mass, total fat and trunk fat mass, as well as visceral adipose tissue mass which will be quantified using Hologic APEX 3.1 software. | 16 weeks
  summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences
Change in physical activity level as assessed using the using the Godin Leisure-Time Exercise Questionnaire. | 16 weeks
  summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences
Change in lipid profile | 16 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences). (total cholesterol: mg/dL; triglycerides: mg/dL; high-density lipoprotein cholesterol mg/dL; low-density lipoprotein cholesterol mg/dL; very low-density lipoprotein cholesterol: mg/dL; cholesterol/HDL ratio mg/dL).
Change in hemoglobin A1c (%) | 16 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences), hemoglobin A1c reported as percentage of average blood sugar level (mg/dL or mmol/L), higher % corresponds to higher average blood sugar levels (normal A1C level is below 5.7%)
Change in c-reactive protein (mg/L) | 16 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences), mg/L (hs-CRP level of 1 mg/L or lower indicates low risk of CVD, hs-CRP level of 1-3 mg/L indicates moderate risk of CVD, hs-CRP level of greater than 3 mg/L indicates high risk of CVD)
Change in interleukin-6 (pg/mL) | 16 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences), pg/mL
Change in tumor necrosis factor alpha (pg/mL) | 16 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences), pg/mL
Change in insulin (mcU/mL) | 16 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences) (mcU/mL)
Change in leptin (ng/mL) | 16 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences) (ng/mL)
Change in adiponectin level (microgram/mL) | 16 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences) (microgram/mL)
Change in insulin-like growth factor (ng/mL) | 16 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences) (ng/mL)
Change in homeostatic model assessment of insulin resistance (estimates beta cell function (%B) and insulin sensitivity (%S), as percentages of a normal reference population) | 16 weeks
  Summarize changes from the baseline to follow-up assessment including calculation of the effect size (mean within-subject difference divided by standard deviation of differences). Plasma glucose: mmol/L (or mg/dL), Insulin: pmol/L (or microunits/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth O'Donnell, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT04220216/ICF_000.pdf